CLINICAL TRIAL: NCT02203903
Title: Multi-institutional Prospective Phase I Research of Expanded Multi-antigen Specifically Oriented Lymphocytes for the Treatment of VEry High Risk Hematopoietic Malignancies
Brief Title: Multi-institutional Prospective Research of Expanded Multi-antigen Specifically Oriented Lymphocytes for the Treatment of VEry High Risk Hematopoietic Malignancies
Acronym: RESOLVE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Collaborators: Children's National Research Institute (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director- Center for Cancer and Immunology Research, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00005533
Record Dates: First submitted 2014-07-25; First posted 2014-07-30 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Relapsed/Refractory Hematopoietic Malignancies, Acute Myeloid Leukemia and MDS
MeSH Terms: conditions — Recurrence; Hematologic Neoplasms; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tumor associated antigen lymphocytes (TAA-T) (Experimental): TAA-T will be infused any time after neutrophil engraftment post-HSCT or day 30, whichever comes first. All infusions will be within 5 months post-HSCT.
  Patients will receive a TAA-T cell dose of 4 x 107 cells/m2.
  Interventions: Biological: Tumor associated antigen lymphocytes (TAA-T)

INTERVENTIONS:
Biological: Tumor associated antigen lymphocytes (TAA-T) — TAA-T may be generated from donors or recipients and will be tested for specificity to 3 tumor antigens commonly found in hematological malignancies (WT1, PRAME, and SURVIVIN,). The goal of this cell infusion will be to initiate an immune response to residual leukemia or lymphoma that includes multiple antigens and may prevent tumor evasion (through decreased expression of a single antigen).

SUMMARY:
This Phase I dose-escalation trial is designed to evaluate the safety of administering rapidly -generated tumor multi-antigen associated -specific cytotoxic T lymphocytes, to HSCT recipients with high risk AML and MDS.

DETAILED DESCRIPTION:
Patients with evidence of high-risk or relapsed or persistent hematopoietic malignancies (for example but not limited to: acute myeloid leukemia and myelodysplastic syndrome (MDS)) will be eligible for this study.

Patients with high risk for relapse will be eligible to receive planned infusion of allogeneic TAA-T after HSCT (with high risk AML and MDS who have undergone allo-HSCT and are in a hematologic remission).

We will utilize our established protocol for the manufacture of tumor multi-antigen associated specific cytotoxic T lymphocytes. Peripheral blood mononuclear cells will be exposed to antigen presenting cells pulsed with peptides to tumor antigens (PRAME, WT1, Survivin) in a cytokine milieu favorable to T cell expansion/activation, inducing selective expansion of T cells targeted to kill tumor cells. Patients would be monitored for the development of toxicity. In patients with disease at the time of TAA-T infusion, efficacy would be evaluated as a secondary endpoint using standard criteria. Exploratory investigational analyses would include monitoring of cytokine and cellular milieu pre- and post- TAA-T infusion and in vitro characterization of the host tumor, donor lymphocyte product, and TAA-T product.

TAA-T will be infused any time after neutrophil engraftment post-HSCT or day 30, whichever comes first at dose level 4 . Infusions will be within first 5 months post-HSCT.

Patients will receive a TAA-T cell dose of 4 x 107 cells/m2.

Each patient will receive at least one infusion according to the enrolled dose level, where the expected volume of infusion is 1 to 10 cc.

If patients with active disease (defined as MRD+ at the time of TAA-T infusion) do not have ≥ grade 3 toxicity that is possibly, probably, or definitely attributed to TAA-T infusion and fail to rapidly progress with disease requiring urgent therapy, patients may receive a subsequent TAA-T cell dose (infusion #2). A subsequent dose (infusion #2) will also be available for those patients who have stable disease or a mixed, partial, or complete response (including continued complete response) by the International Working Group (IWG) criteria (see section 4.2.1) at the evaluation after the first TAA-T infusion.

Patients who have received at least 2 infusions of TAA-T are eligible to receive up to 6 additional doses (infusion #3 to #8) of TAA-T at monthly intervals each of which will consist of the same cell number as their enrolled dose level. Patients will not be able to receive additional doses until the initial safety profile is completed at 28 days following the second infusion. Notably, these doses will be identical to the treated dose for this patient (i.e. no subsequent dose escalation). Patients would then receive additional doses starting greater than 28 days from second infusion and be treated at the same dose level as he/she has previously received.

ELIGIBILITY:
Recipient Inclusion Criteria to Enter Protocol:

* Aged 6 months to 80 years.
* Anticipated myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant.
* Patients with high risk AML and MDS who have received or will receive an allo-HSCT and have not had hematologic relapse of disease.
* Karnofsky/Lansky score of ≥ 50.
* Agree to use contraceptive measures during study protocol participation (when age appropriate).
* Patient or parent/guardian capable of providing informed consent.
* T cell chimerism > 94% if collected from recipient of allo-HSCT

Recipient Exclusion Criteria to Enter Protocol:

* Patients with uncontrolled infections.
* Current evidence of GVHD > grade 2 or bronchiolitis obliterans syndrome, sclerotic GVHD, or serositis.
* Pregnancy (female of childbearing potential).

Recipient Inclusion Criteria for TAA-T Administration:

* Patients with high risk AML and MDS who have received an allo-HSCT and have not had hematologic relapse of disease.
* Steroids less than 0.5 mg/kg/day prednisone or equivalent in the context of no escalation of treatment within the preceding 2 weeks
* Karnofsky/Lansky score of ≥ 50.
* Bilirubin < 2.5 mg/dL, AST/ALT <5x upper limit of normal, Serum creatinine < 1.0 or 2x the upper limit of normal (whichever is higher).
* Pulse oximetry of > 90% on room air.
* Absolute neutrophil count > 250/ µL (may be supported with Granulocyte colony-stimulating factor (GCSF)).
* Agree to use contraceptive measures during study protocol participation (when age appropriate).
* Patient or parent/guardian capable of providing informed consent.
* LVEF > 50% or LVSF > 27% (performed within the last 6 months) if history of TBI >500 cGy for arm A and B.
* Total chimerism > 50%; or if cancer cells preclude this, donor T cell chimerism > 50% (performed within the last 6 months).

Recipient Exclusion Criteria for TAA-T Administration:

* Patients who received ATG, Campath, or other T cell immunosuppressive monoclonal antibodies within 28 days prior to TAA-T infusion.
* No investigational therapies (under IND, not extensively studied in the current clinical context) within 28 days prior to TAA-T infusion.
* Uncontrolled infections.
* Active Bronchiolitis obliterans syndrome, sclerotic GVHD, or serositis.
* Active acute GVHD or chronic GVHD requiring escalation of treatment within preceding 2 weeks of any grade is exclusion for Arm C patients.
* Pregnancy or lactating (female of childbearing potential).
* Patients who have or will be receiving 2nd allogeneic HSCT

Donor Inclusion Criteria:

* Donors for allogeneic (i.e. HLA matched or mismatched related or unrelated) stem cell transplants who have undergone eligibility evaluation as per FDA regulations outlined in 21 CFR 1271 subpart C. If a donor has been chosen for the transplant based on urgent medical need, that same donor will also be used for TAA-T generation provided that there are no new reasons for ineligibility since the transplant donor evaluation.
* Aged 6 months to 80 years.
* Donor or guardian of pediatric capable of providing informed consent.
* Donor must have completed infectious Disease (ID) testing up to 7 days before or after the collection of blood from the donor (related or unrelated) for TAA-T manufacturing. The following tests will be performed:

  * HBsAg
  * HB Core antibody
  * HIV1/2 NAT
  * Syphilis (T. Pallidum IgG)
  * HTLV I/II
  * CMV total
  * HBV/HCV NAT
  * West Nile Virus NAT.
  * Cruz (Chagas) antibody
  * Hepatitis C
* Female donors of childbearing age must have a negative pregnancy test within 7 days of blood collection for TAA-T manufacturing.

Donor Exclusion Criteria:

* Donation of cells would pose a physical or psychological risk to the donor.
* Female donors of childbearing age who are known to be pregnant.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
Safety of investigational product (TAA-T) | 45 days
  Acute GVHD grades III-IV within 45 days of the last dose of TAA-T
Safety of TAA-T cells | 45 days
  Grades 3-5 infusion-related adverse events within 45 days of the last dose of TAA-T
Safety of TAA-Ts | 45 days
  Grades 4-5 non-hematological attributable adverse events within 45 days of TAA-T dose and that are not due to the pre-existing infection or the original malignancy or pre-existing co-morbidities as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0
Event-free survival | Twelve months post-HSCT
  To determine if event-free survival (EFS) at twelve months post-HSCT is improved with TAA-T administration for AML and MDS (Arm C).

SECONDARY OUTCOMES:
Tumor associated antigen lymphocytes (TAA-T) responses | 2 years
  To determine the number of patients who respond to tumor multi-antigen associated specific cytotoxic lymphocytes (TAA-T) for treatment for high risk or relapsed or refractory hematopoietic malignancies as defined by those who maintain or achieve CR, PR, MR or SD following TAA-T infusion and evaluate if this was associated with in vivo persistence of TAA-T

OTHER OUTCOMES:
The incidence and severity of acute and/or chronic GVHD | 2 years
  To determine the incidence and severity of acute and/or chronic GVHD in patients treated with TAA-T and compare this to historical controls
Event free and overall survival | 1 year
  Event free and overall survival at 1 year for patients enrolled under Arm C.
Characterize the cytokine and lymphocyte cellular milieu pre- and post-infusion of TAA-T | 2 years
  To characterize the cytokine and lymphocyte cellular milieu pre- and post-infusion of TAAT in vivo.
Compare specificity to tumor antigens before and after TAA-T infusion | 2 years
  To characterize the TAA-T generated prior to infusion in terms of specificity to tumor antigens and compare this with tumor antigens present on patient samples, evaluating for in vitro activity of TAA-T.
To evaluate the incidence of post-transplant complications after TAA-T infusion. | 45 days
  To evaluate the incidence of other post-transplant complications such as engraftment, sinusoidal obstructive syndrome, neutropenia and significant infections during the period of monitoring after cellular infusion.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Tania Jain, MD, Baltimore, Maryland

REFERENCES:
- [Derived] Kinoshita H, Cooke KR, Grant M, Stanojevic M, Cruz CR, Keller M, Fortiz MF, Hoq F, Lang H, Barrett AJ, Liang H, Tanna J, Zhang N, Shibli A, Datar A, Fulton K, Kukadiya D, Zhang A, Williams KM, Dave H, Dome JS, Jacobsohn D, Hanley PJ, Jones RJ, Bollard CM. Outcome of donor-derived TAA-T cell therapy in patients with high-risk or relapsed acute leukemia post allogeneic BMT. Blood Adv. 2022 Apr 26;6(8):2520-2534. doi: 10.1182/bloodadvances.2021006831. PMID 35244681